CLINICAL TRIAL: NCT01076712
Title: The Effectiveness of Physiotherapy Interventions in Patients With Parkinson's Disease, a Randomized Controlled Trial
Brief Title: Effectiveness of Physiotherapy Interventions for Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: WOO Cheuk Wai, Physiotherapy Department, Queen Elizabeth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCKESOP0016a
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Prenatal Education; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy Interventions (Experimental): Physiotherapy Interventions including strengthening exercise, balance training, gait training with visual cue, gait training with treadmill.
  Interventions: Other: Physiotherapy Interventions
- Education (Other): Education
  Interventions: Other: Education Classes

INTERVENTIONS:
Other: Physiotherapy Interventions — Physiotherapy interventions including strengthening exercise, balance training, gait training with visual cus and gait training with treadmill
  Arms: Physiotherapy Interventions
Other: Education Classes — Education Classes
  Other Names: Education
  Arms: Education

SUMMARY:
Parkinson's Disease is an incurable and progressive disease. Treatment includes medication and non-pharmacological intervention such as physiotherapy. Physiotherapy is a main component of non-pharmacological interventions. It includes exercise to strengthen the muscles; improves balance and walking, and adopts the use of visual cue training. Treatment has been found to be effective in patients with mild impairment up to 6 months post-treatment. The present study will investigate the effectiveness of treatment for patients with mild to moderate impairment for short term (3-month) and long term (1 year). The hypothesis is that compared to patient education alone, physiotherapy intervention for patients with Parkinson's disease leads to improve function and quality of life.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is an incurable and progressive disease (Rubenis 2007). Current management include medical, neuro-surgical and non-pharmacological intervention. Physiotherapy is a major component in non-pharmacological interventions. Effective interventions including visual or auditory cues improves gait (Nieuwboer et al. 2007), exercise is effective in improving balance (Hirsch et al 2003); intense treadmill training improves motor control, quality of life and walking speed so as to sustain improvement in gait speed and motor control post 4 weeks of treatment (Herman et al 2007). Patient with PD attending physiotherapy twice weekly, one and half hour for 12 weeks showed improvement in walking speed and Activities of Daily Living (Ellis et al 2005). However, the majority of focus on patients in the Hoehn and Yahr stage of 2 to 3 and long term effect is lacking (Kwakkel et al 2007). A knowledge gap is present in the effectiveness of physiotherapy training of patients with Parkinson's disease in the more advanced stage of disease and long term effect is lacking. The aim of the study is to investigate the immediate, short-term & long-term clinical effects of physiotherapy training of patients with Parkinson's disease. The hypothesis is that compared to patient education alone, physiotherapy intervention for patients with Parkinson's disease leads to improve function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Stable medication usage
* Hoehn and Yahr stage II to IV
* At least 1 score of 2 or more for at least 1 limb of either the tremor, rigidity, or bradykinesia item of the Unified Parkinson's Disease Rating Scale (UPDRS)
* Able to walk independently
* No severe cognitive impairments (Mini-Mental State Examination - Chinese Cantonese version) score greater than 24

Exclusion Criteria:

* Other severe neurological, cardiopulmonary, or orthopedic disorders
* Having participated in a physiotherapy or rehabilitation program in previous 2 months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention
Levodopa equivalent daily dosage (LEDD) | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention

SECONDARY OUTCOMES:
Timed Up and Go Test | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention
Activities-Specific Balance Confidence Scale (Chinese version) | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention
Parkinson's Disease Questionnaire (Standard Chinese Version) | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention
  Parkinson's Disease Questionnaire (Standard Chinese Version) - PDQ-39 (Chinese)
Number of Injurious Falls | Baseline. Immediate, 3-month, 6-month and 1 year Post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: CW WOO, Principal Investigator — Physiotherapy Department, Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

REFERENCES:
- [Background] Nieuwboer A, Kwakkel G, Rochester L, Jones D, van Wegen E, Willems AM, Chavret F, Hetherington V, Baker K, Lim I. Cueing training in the home improves gait-related mobility in Parkinson's disease: the RESCUE trial. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):134-40. doi: 10.1136/jnnp.200X.097923. PMID 17229744
- [Background] Hirsch MA, Toole T, Maitland CG, Rider RA. The effects of balance training and high-intensity resistance training on persons with idiopathic Parkinson's disease. Arch Phys Med Rehabil. 2003 Aug;84(8):1109-17. doi: 10.1016/s0003-9993(03)00046-7. PMID 12917847
- [Background] Herman T, Giladi N, Gruendlinger L, Hausdorff JM. Six weeks of intensive treadmill training improves gait and quality of life in patients with Parkinson's disease: a pilot study. Arch Phys Med Rehabil. 2007 Sep;88(9):1154-8. doi: 10.1016/j.apmr.2007.05.015. PMID 17826461
- [Result] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Result] Morris S, Morris ME, Iansek R. Reliability of measurements obtained with the Timed "Up & Go" test in people with Parkinson disease. Phys Ther. 2001 Feb;81(2):810-8. doi: 10.1093/ptj/81.2.810. PMID 11175678
- [Result] Mak MK, Lau AL, Law FS, Cheung CC, Wong IS. Validation of the Chinese translated Activities-Specific Balance Confidence scale. Arch Phys Med Rehabil. 2007 Apr;88(4):496-503. doi: 10.1016/j.apmr.2007.01.018. PMID 17398252
- [Result] Tsang KL, Chi I, Ho SL, Lou VW, Lee TM, Chu LW. Translation and validation of the standard Chinese version of PDQ-39: a quality-of-life measure for patients with Parkinson's disease. Mov Disord. 2002 Sep;17(5):1036-40. doi: 10.1002/mds.10249. PMID 12360555
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886